CLINICAL TRIAL: NCT07354672
Title: Pathogen-Reduced Platelet Concentrates: Experience In Routine Practice In Germany
Acronym: INITIATE
Status: Recruiting | Type: Observational
Sponsor: Deutsches Rotes Kreuz DRK-Blutspendedienst Baden-Wurttemberg-Hessen (Other)
Responsible Party: Sponsor
Other Study IDs: INITIATE
Record Dates: First submitted 2025-11-26; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Platelet Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Pathogen-Reduced Platelet Concentrates — Pathogen-reduced platelet concentrates which were either produced from 4, 5 or 8 buffy coats from whole blood donations or which were collected by apheresis.

SUMMARY:
* Overall objective: to accumulate further experience with the use of pathogen-reduced platelet concentrates throughout the entire process chain from manufacture to clinical use of pathogen-reduced platelet concentrates and their efficacy and safety under real-world conditions. The study aims to better understand the impact of pathogen inactivation on the various steps of the overall supply chain in routine practice, whereby safety, measured in terms of the frequency of serious transfusion reactions and the type, imputability, and outcome of the reactions, is the primary endpoint.
* Study product: Pathogen-reduced platelet concentrates.
* Methodology: multi-center, open-label, prospective, non-interventional safety study.

DETAILED DESCRIPTION:
The safety of blood products has significantly improved over the past 30 years due to enhanced donor selection and more sensitive testing for infectious agents. Nevertheless, a residual risk remains, particularly the risk of bacterial contamination in platelet concentrates. To mitigate this, pathogen reduction methods and/or bacterial detection tests can be employed. In Germany, there is currently limited large-scale experience under real-world conditions regarding how pathogen reduction of platelet concentrates (PC) affects the various stages of the process chain from production, distribution through to the clinical application and its impact on safety and efficacy.To better understand the effects, the non-interventional post-authorization safety study INITIATE evaluates various aspects of pathogen-reduced, platelet concentrates across the entire process chain and compares results to historical data of standard, non-pathogen reduced PC. This project is a multi-center, open-label, prospective, non-interventional post-authorisation safety-study and is divided into two parts:

Part 1 focuses on product- and process-related objectives. It includes all pathogen-reduced PC units produced at participating manufacturing sites to analyse the product and supply-related endpoints including manufacturing data, quality control data, logistics and supply, safety and costs. Part 1 shall include data on 20.000 PC.

Part 2 includes a defined number of patients requiring PC transfusions at participating clinical study centers. It aims to collect data on safety (primary and co-primary endpoint: transfusion reactions (frequency, type, severity, imputability and outcome, according to CTCAE) and efficacy (bleeding, platelet increment (subgroup of patients), alloimmunization or platelet refractoriness). Part 2 shall include 850 patients (with an expected total number of 4.500 to 5.000 PC transfusions).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients who, based on clinical indications*, receive at least one platelet transfusion with a pathogen-reduced platelet concentrate for treatment of bleeding risk caused by severe thrombocytopenia resulting from impaired platelet production.

(* Taking into account the Cross-sectional Guidelines on the transfusion of blood components and plasma derivatives issued by the German Medical Association (Bundesärztekammer) in its current version.)

Exclusion Criteria:

Patients will not be included if they fulfil at least one of the following exclusion criteria:

* Known hypersensitivity to amotosalen HCl or psoralens. In this case, platelet concentrates treated with this pathogen inactivation method should not be used.
* Known allergies of the recipient to human plasma proteins.
* Known immune thrombocytopenia.
* Thrombotic microangiopathy (thrombotic thrombocytopenic purpura; haemolytic uremic syn-drome).
* Post-transfusion purpura.
* Heparin-induced thrombocytopenia.
* Congenital platelet function disorders, such as Glanzmann's thrombasthenia or Bernard- Souli-er syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who, based on clinical indications*, receive at least one platelet transfusion with a pathogen-reduced platelet concentrate for treatment of bleeding risk caused by severe thrombocytopenia resulting from impaired platelet production.
  (* Taking into account the Cross-sectional Guidelines on the transfusion of blood components and plasma derivatives issued by the German Medical Association (Bundesärztekammer) in its current version.)
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of serious transfusion reactions after transfusion of pathogen-reduced platelet concentrates | Within 24 hours (acute) and up to 6 weeks (delayed) depending on transfusion reaction
Type, imputability and outcome of serious adverse reactions after transfusion of pathogen-reduced platelet concentrates. | Within 24 hours (acute) and up to 6 weeks (delayed) depending on transfusion reaction

SECONDARY OUTCOMES:
Number of severe bleeding events | Within 24 hours after platelet transfusion
  Number of severe bleeding events per patient
Frequency of severe bleeding events | Within 24 hours after platelet transfusion
  Proportion of patients with at least one severe bleeding event
Clinical outcome of severe bleeding events | Through study completion, up to 18 months
  Outcome categorized as resolved, ongoing, or fatal
Overall survival | From date of enrollment until date of death from any cause, assessed up to 18 months
  Time-to-event analysis of overall survival
Cause of death | From date of enrollment until date of death from any cause, assessed up to 18 months.
  Categorized cause of death
Daily number of pathogen-reduced platelet concentrates manufactured | Through study completion, up to 18 months
  Number of pathogen-reduced platelet concentrates manufactured per day
Manufacturing Workload for Pathogen-Reduced Platelet Concentrates | Through study completion, up to 18 months
  Cumulative hands-on manufacturing time per product
Manufacturing duration of pathogen-reduced platelet concentrates | Through study completion, up to 18 months
  Time from start to completion of manufacturing
Manufacturing failure rate | through study completion, up to 18 months
  Number and proportion of manufacturing failures
Availability of platelet concentrates for supply | Through study completion, up to 18 months
  Number of released platelet concentrates available for distribution
Time from product release to distribution | Through study completion, up to 18 months
  Time from release of platelet concentrates to transfer to the distribution department
Shelf-life extension of non-pathogen-reduced platelet concentrates | Through study completion, up to 18 months
  Number of non-pathogen-inactivated platelet concentrates requiring shelf-life extension
Discard rate of platelet concentrates | Through study completion, up to 18 months
  Number of platelet concentrates discarded
Platelet content of pathogen-reduced platelet concentrates | Through study completion, up to 18 months
  Platelet content per pathogen-reduced platelet concentrate
Bacterial contamination of pathogen-reduced platelet concentrates | Through study completion, up to 18 months
  Presence or absence of baterial contamination per platelet concentrates as determined by routine quality control testing
pH of pathogen-reduced platelet concentrats at end of sheld life | Through study completion, up to 18 months
  pH value measured at the end of shelf life
Residual leukocyte count | Through study completion, up to 18 months
  Residual leukocyte count per platelet concentrate
Out-of-Specification platelet concentrates | Through study completion, up to 18 months
  Proportion of platelet concentrates outside of predefined quality specifications
Transfusion reactions | Within 24 hours (acute) and up to 6 weeks (delayed) depending on transfusion reaction
  Number of acute and delayed transfusion reactions
HLA Alloimmunisation | Through study completion, up to 18 months
  Incidence of newly detected HLA antibodies
Composite thrombelastographhy coagulation index | at least one measurement between 10 minutes and 24 hours post transfusion
  Composite index derived from predefined thrombelastography parameters
Fibrinogen concentration | at least one measurement between 10 minutes and 24 hours post transfusion
  Change in fibrinogen concentration after platelet transfusion
Time to next platelet concentrate transfusion under routine conditions | From completion of first transfusion until the next transfusion under routine clinical practice, assessed up to 18 months
  Time interval to subsequent platelet transfusion
Number of platelet concentrates per patient | through study completion, up to 18 months
  Total number of platelet transfusions per patients
Number of Red Blood Cell Transfusions per patient | Through study completion, up to 18 months
  Total number of packed red blood cell transfusions per patient.
Number of Plasma Transfusions per patient | Through study completion, up to 18 months
  Total number of plasma transfusions per patient
Cost of Platelet Concentrate products | through study completion, up to 18 months
  Direct costs of platelet concentrate products
Reimbursement of platelet concentrates within the DRG System | Through study completion, up to 18 months
  Reimbursement of platelet concentrates by health insurance providers
User satisfaction at the various stages of production, distribution and application of platelet concentrates | Through study completion, up to 18 months
  User satisfaction at the various stages of production, distribution and application of platelet concentrates, measured on a scale of 0 to 10, with 10 representing best result, based on questionnaires at the start of the observational study, after three and six months and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Schrezenmeier, Prof. Dr. med., Study Director — Institut für Klinische Transfusionsmedizin und Immungenetik Ulm gGmbH (DRK-Blutspendedienst Baden-Württemberg Hessen gGmbH und Universitätsklinikum Ulm AöR). Institut für Transfusionsmedizin, Universität Ulm
Locations (1):
- Institut für Klinische Transfusionsmedizin (IKT) und DRK Blutspendedienst Baden-Württemberg-Hessen/ Transfusionsambulanz MVZ DRK-Blutspendedienst Ulm gGmbH, Ulm, Baden-Wurttemberg, Germany